CLINICAL TRIAL: NCT03989063
Title: Motor Learning in Individuals With Lower Limb Loss and Chronic Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nevada, Las Vegas (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 1299365; 1K01HD091449-01A1 (NIH)
Record Dates: First submitted 2019-06-04; First posted 2019-06-18 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Amputation; Diabetes Mellitus; Neuropathy, Diabetic
Keywords: Motor Learning; Attentional Focus; Limb Loss; Diabetes; Balance
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Neuropathies

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of the two conditions receiving either external or internal attentional focus instructions for the same balance task. After a washout period of at least 1 month, the participant will repeat the experiment with instruction not previously received (i.e. if the participant received the internal focus instruction during the first phase, he/she will receive the external focus instruction in the second phase).
Who Masked: Participant
Masking Description: Participants are randomly assigned to one of the two parallel groups receiving either external or internal attentional focus instructions for the same balance task. Participants will be blinded to this group assignment until final debriefing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Amputees (External Focus) (Experimental): Participants in this group will receive the external focus instruction on where to direct their attention while training to perform the balance task. During training, the assigned instruction will be reinforced at the beginning and after every 5 practice trials.
  Interventions: Behavioral: Instructions to perform a motor task (external vs. internal focus instructions)
- Amputees (Internal Focus) (Active Comparator): Participants in this group will receive the internal focus instruction on where to direct their attention while training to perform the balance task. During training, the assigned instruction will be reinforced at the beginning and after every 5 practice trials.
  Interventions: Behavioral: Instructions to perform a motor task (external vs. internal focus instructions)
- Diabetes (External Focus) (Experimental): Participants in this group will receive the external focus instruction on where to direct their attention while training to perform the balance task. During training, the assigned instruction will be reinforced at the beginning and after every 5 practice trials.
  Interventions: Behavioral: Instructions to perform a motor task (external vs. internal focus instructions)
- Diabetes (Internal Focus) (Active Comparator): Participants in this group will receive the internal focus instruction on where to direct their attention while training to perform the balance task. During training, the assigned instruction will be reinforced at the beginning and after every 5 practice trials.
  Interventions: Behavioral: Instructions to perform a motor task (external vs. internal focus instructions)

INTERVENTIONS:
Behavioral: Instructions to perform a motor task (external vs. internal focus instructions) — During the balance task, the participants will receive instructions to focus on external targets (external focus group) vs. movement of the body (internal focus group).

SUMMARY:
Inadequate rehabilitation training after amputation can result in poor patient outcomes, injuries, and wasted healthcare resources. This is a serious public health problem due to an aging population and rising prevalence of diabetes (main cause of amputation in the U.S.). In this study, the investigators will examine the effects of external vs. internal attentional focus instruction on learning of a balance task in individuals with existing amputation and those at risk of amputation (older adults with diabetes). With the proposed research, the investigators aim to expand the understanding of motor learning in individuals with and at risk of lower limb loss to provide knowledge that will lead to more effective and efficient rehabilitation.

DETAILED DESCRIPTION:
1. Prior to participation in the study, the purpose and procedures of the study, including possible image and video recordings, will be explained to the subjects.
2. Subjects will then be required to give written consent for their participation and will receive a copy of their consent form.
3. The following 2-part research protocol uses a similar experimental protocol (learning a balance task) on individuals with leg amputation (Part 1), and individuals with chronic diabetes (Part 2).

Part 1:

The experiment will take place over a 3-day period including screening and baseline testing (Visit 1), balance training (Visits 2), and retention testing (Visit 3; at least 24 hours after Visit 2). On Visit 1, the investigators will assess aspects of health and functional capacity to assess participation eligibility and establish baseline characteristics of the participants. In addition to medical history and anthropometric measurements, the assessment will consist of clinical surveys of quality of life, physical activity level, balance confidence, and fear of falling. Ambulatory performance will be quantified. Additional amputee-specific measures will be used to assess functional characteristics unique to the population.

The balance training involves standing and maintaining balance on a stabilometer, which consists of a platform (1.3m long by 1.4m wide) connected to a single axis that allows bi-directional sway (Lafayette Instrument Co.; Figure 1). The maximum angular deviation of the platform is 18°. A safety harness is provided to prevent falls but does not provide support during the performance of the task. The load on the harness will be monitored with an S-type strain gauge (Delsys Inc., Massachusetts, USA) connected in series to the harness tether. Participants are required to maintain balance with feet in a medial-lateral orientation while standing on the balance board and looking straight ahead. A potentiometer monitors the sway angle of the platform. An integrated timer measures time in balance, which is defined as when the platform angle is within ± 5° of horizontal.[52] The primary outcome measure is time in balance (sec.) for each 30s trial. The secondary outcome measure is platform angular deviation from horizontal (RMSE; degree).

Participants will be assigned to receive the 2 attentional focus conditions in random order. Depending on the condition, participants will receive either internal or the external focus instruction on where to direct their attention while training to perform the balance task. During training, the assigned instruction will be reinforced at the beginning and after every 5 practice trials. After they complete training with the first condition, they will go through a washout period (at least 4 weeks) before receiving training under the other condition. Participants will be blinded to the purpose of the intervention and study design until debriefing at the end of the study.

The training will take place over a 2-day period (Visits 1 and 2), the investigators will monitor the changes in balance task performance over 40 total practice trials (20 trials each visit). The balance training consists of thirty 30s trials with a 90s rest interval between trials. During the rest interval, the platform will be locked to provide a stable surface or the participant can choose to step off the platform to sit down and rest when needed. After each 5 trials, participants will be given feedback regarding their performance (time in balance). No additional feedback will be provided. This protocol has been validated in the older adult population (mean age 69.4 years) in a previous study (Chiviacowsky et al. 2010). After each training block of 5 trials, the participant's self-perceived direction of attentional focus and spontaneous comments during the practice will be checked. The retention test will be performed at least 24 hours after the 2nd training day (Visit 3). The retention test will consist of performing 10 trials of the same balance task during which the participant will not receive any instructions, reminders, or feedback. An additional 10 trials of skill transfer task will be performed with an added cognitive task (counting numbers backward).

Part 2 (individuals with diabetes):

The procedure of Part 2 of this research is identical to Part 1. The main differences, in addition to the different participant population are described below.

In addition to the baseline health and functional capacity assessments as described in Part 1, the investigators will assess all participants' sensorimotor function using an established knee joint reposition sense test on a Cybex Norm dynamometer (Computer Sports Medicine Inc., Stoughton, MA, USA). This test assesses participant's ability to reproduce a joint angle using only proprioception. The test performance will be measured as the absolute error in degrees between the reproduced and target angles. This specific test was chosen to quantify the lower limb sensorimotor function because previous studies have shown it to be predictive of mobility outcomes in older adults in general and in those with diabetes. The investigators will determine individuals with diabetes-related sensorimotor impairment if the error is greater than 3.65°.

Individuals will be randomly assigned to receive either internal or external focus instructions conditions during the balance training. The experimental protocols and procedures will be the same as in Aim 1, including the screening (Visit 1), balance training (Visits 2), and retention and skill transfer testing (Visit 3; at least 24 hours after Visit 2).

ELIGIBILITY:
Inclusion Criteria (amputees):

1. Have unilateral transtibial or transfemoral amputation,
2. Age >18 years,
3. Are fitted with a walking prosthesis and use it regularly and proficiently (K-level of 2 or above, further defined as scoring higher than 50 percentile on the Prosthetic Limb Users Survey of Mobility),
4. Able to stand for at least 5 minutes without using an assistive device or experiencing excessive fatigue
5. Willing to travel to UNLV 6 times for training and testing.

The inclusion criteria (non-amputee older adults with and without chronic diabetes):

1. Age >18 years,
2. With or without a current diagnosis of type II diabetes
3. Able to walk for at least 50 meters without assistance from other people,
4. Able to stand for at least 5 minutes without using an assistive device or experiencing excessive fatigue
5. Willing to travel to UNLV 6 times for training and testing. -

Exclusion Criteria:

1. Have other concurrent central nervous system diseases that influence motor functions and balance.
2. Have leg/foot ulcer or other conditions that cause pain during weight-bearing.
3. Have cardiovascular, respiratory or other critical health conditions that preclude moderate physical activity.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in balance performance | Throughout the training period (2 days, up to 40 trials) and during the post-training tests
  During each 30-second balance practice trial, time in balance which is defined as when the balance platform is within 5 degrees from horizontal will be measured in seconds. A longer time in balance (up to 30 seconds) indicates better balance performance.
Change in balance performance | Throughout the balance training period (2 days, up to 40 trials) and during the post-training tests
  During each balance practice trial, average deviation of balance platform angle from horizontal will be measured in degrees. Smaller deviation from horizontal indicates better balance performance.

SECONDARY OUTCOMES:
Change in fall recovery performance | Before and after balance training. The after training assessment will be conducted 2-10 days after the conclusion of the balance training.
  Rate of successful recovery from 10 trials of simulated tripping/slipping perturbation during walking on a treadmill will be measured in percentage. Higher percentage of successful recovery indicates better fall recovery performance.
Change in fall recovery performance | Before and after the 2-day balance training. The after training assessment will be conducted 2-10 days after the conclusion of the balance training.
  Trunk flexion angle during slipping/tripping (degrees). Previous studies have shown that smaller trunk angle during simulated tripping/slipping is associated with successful fall recovery. Smaller trunk flexion angle indicates better fall recovery performance.
Change in fall recovery performance | Before and after the 2-day balance training. The after training assessment will be conducted 2-10 days after the conclusion of the balance training.
  Trunk angular velocity during slipping/tripping (degree/second). Previous studies have shown that slower trunk angle change (i.e. lower trunk angular velocity) during simulated tripping/slipping is associated with successful fall recovery. Slower trunk angular velocity indicates better fall recovery performance.
Change in patient's self-reported outcomes | Throughout the balance training period (2 days, assessed every 5 practice trials).
  Self-efficacy regarding the performance of the balance task is assessed using a 4-question survey. An example question is: "How confident are you that you can keep yourself in balance for 15 out of 30 seconds?". Participant's response to each question is measured using a 0-10 scale. Higher confidence indicates greater self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Szu-Ping Lee, PhD, Principal Investigator — University of Nevada, Las Vegas
Locations (1):
- University of Nevada, Las Vegas, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) collected in this study is specific to the study protocol only. Sharing of the IPD to other researchers would pose a risk to participant privacy, and is not scientifically merited.

REFERENCES:
- [Background] Chiviacowsky S, Wulf G, Wally R. An external focus of attention enhances balance learning in older adults. Gait Posture. 2010 Oct;32(4):572-5. doi: 10.1016/j.gaitpost.2010.08.004. Epub 2010 Sep 17. PMID 20850325

DOCUMENTS (2):
  • Informed Consent Form: For participants with diabetes (study part 2) (2021-04-26): https://cdn.clinicaltrials.gov/large-docs/63/NCT03989063/ICF_002.pdf
  • Informed Consent Form: For participants with amputation (study part 1) (2021-04-26): https://cdn.clinicaltrials.gov/large-docs/63/NCT03989063/ICF_003.pdf